CLINICAL TRIAL: NCT01462344
Title: A 6-month Safety and Benefit Study of Inhaled Fluticasone Propionate/ Salmeterol Combination Versus Inhaled Fluticasone Propionate in the Treatment of 6,200 Pediatric Subjects 4-11 Years Old With Persistent Asthma
Brief Title: 6-month Safety and Benefit Study of ADVAIR in Children 4-11 Years Old
Acronym: VESTRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115358
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: pediatric; ADVAIR; FLOVENT; asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ADVAIR 100/50mcg (Experimental): fluticasone propionate/salmeterol combination (100/50mcg) twice daily (AM and PM) for 6 months
  Interventions: Drug: ADVAIR 100/50mcg
- ADVAIR 250/50mcg (Experimental): fluticasone propionate/salmeterol combination (250/50mcg) twice daily (AM and PM) for 6 months
  Interventions: Drug: ADVAIR 250/50mcg
- FLOVENT 100mcg (Active Comparator): fluticasone propionate (100) twice daily (AM and PM) for 6 months
  Interventions: Drug: FLOVENT 100mcg
- FLOVENT 250mcg (Active Comparator): fluticasone propionate (250mcg) twice daily (AM and PM) for 6 months
  Interventions: Drug: FLOVENT 250mcg

INTERVENTIONS:
Drug: ADVAIR 100/50mcg — fluticasone propionate/salmeterol combination (100/50mcg) twice daily (AM and PM) for 6 months
  Other Names: FSC 100/50
  Arms: ADVAIR 100/50mcg
Drug: ADVAIR 250/50mcg — fluticasone propionate/salmeterol combination (250/50mcg) twice daily (AM and PM) for 6 months
  Other Names: FSC 250/50
  Arms: ADVAIR 250/50mcg
Drug: FLOVENT 100mcg — fluticasone propionate (100) twice daily (AM and PM) for 6 months
  Other Names: FP 100
  Arms: FLOVENT 100mcg
Drug: FLOVENT 250mcg — fluticasone propionate (250mcg) twice daily (AM and PM) for 6 months
  Other Names: FP 250
  Arms: FLOVENT 250mcg

SUMMARY:
The purpose of this study is to assess whether the risk of serious asthma-related events (asthma-related hospitalizations, endotracheal intubations, and deaths) in children 4-11 years old taking inhaled fluticasone propionate/salmeterol combination is the same as those taking inhaled fluticasone propionate alone.

DETAILED DESCRIPTION:
Progress of Enrollment, Updated Annually: This study has been completed and the final clinical study report was submitted to the FDA in May of 2016. This is the final update, as this study is complete.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in the study
2. Age 4-11 years old
3. Male or eligible female - Female subjects should not be enrolled if they are pregnant, lactating or plan to become pregnant during the time of study participation
4. Asthma diagnosis for at least 6 months
5. Ability to answer questions regarding asthma control and use a metered dose inhaler and DISKUS
6. A history of clinical varicella infection or recipient of a varicella vaccine in countries where the product label includes a warning regarding more serious chickenpox infections in patients using corticosteroids.
7. History of at least once occurrence of asthma exacerbation within the prior 12 months
8. Currently being treated for asthma and no change in asthma therapy for the last 4 weeks (Eligible subjects include: subjects with use of short-acting beta-agonist, leukotriene receptor antagonist, theophylline, or cromolyn whose asthma is not well-controlled; subjects on low-dose ICS monotherapy whose asthma is not well-controlled; subjects on low-dose ICS and one or more adjunctive therapy whose asthma is either controlled or not well-controlled asthma; subjects on medium-dose ICS monotherapy whose asthma is either controlled or not well-controlled; and subjects on medium-dose ICS and one or more adjunctive therapy whose asthma is well-controlled)

Exclusion Criteria:

1. History of life-threatening asthma
2. Unstable asthma
3. Current use of high-dose ICS or ICS/LABA therapy to treat asthma symptoms
4. Concurrent respiratory disease: Current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, allergic bronchopulmonary aspergillosis, cystic fibrosis, bronchopulmonary dysplasia, or other severe respiratory abnormalities other than asthma.
5. Respiratory infection
6. Subjects with only exercise-induced asthma
7. An asthma exacerbation within the last 4 weeks or more than 4 separate exacerbations in the last 12 months
8. Hospitalization for asthma within 4 weeks or more than 2 hospitalizations within the last 12 months
9. Other current evidence of clinically significant uncontrolled disease/conditions of any body or organ system
10. Neurological or psychiatric disease or history of drug or alcohol abuse of a subject or his/her guardian which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirements
11. Participation in an interventional study or used any investigational drug for any disease state within the last 30 days
12. Any adverse reaction including immediate or delayed hypersensitivity to any beta-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy, or vehicle contained within these medication
13. Severe hypersensitivity to cow's milk proteins
14. Administration of prescription or over the counter medications that would significantly affect the course of asthma, or interact with sympathomimetic amines such as: anti-IgE (omalizumab), anticonvulsants (barbiturates, hydantoins, carbamazepine); polycyclic antidepressants, beta-adrenergic blockers; phenothiazines, monoamine oxidase inhibitors, or diuretics
15. Potent cytochrome P450 3A4 (CYP3A4) inhibitors within the last 4 weeks (e.g., ritonavir, ketoconazole, itraconzole)
16. Affiliation with investigator's site, including a immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
17. A Child in Care (CiC) is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6250 (Actual)
Dates: Start 2011-11-17; Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (425):
- United States (211):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Scottsboro, Alabama
  - GSK Investigational Site, Toney, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Dothan, Alaska
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bentonville, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Alhambra, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Canoga Park, California
  - GSK Investigational Site, Dinuba, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Gold River, California
  - GSK Investigational Site, Granada Hills, California
  - GSK Investigational Site, Harbor City, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Napa, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Est., California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Marino, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, West Sacramento, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Destin, Florida
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pace, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Ponte Vedra Beach, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Calhoun, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Shiloh, Illinois
  - GSK Investigational Site, Crown Point, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Largo, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, White Marsh, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Buckley, Michigan
  - GSK Investigational Site, Fenton, Michigan
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Port Gibson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Livingston, New Jersey
  - GSK Investigational Site, Marlton, New Jersey
  - GSK Investigational Site, Northfield, New Jersey
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Somerville, New Jersey
  - GSK Investigational Site, Verona, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Astoria, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Newburgh, New York
  - GSK Investigational Site, North Syracuse, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Westfield, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Beavercreek, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Marion, Ohio
  - GSK Investigational Site, Shaker Heights, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Wheeling, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Belle Vernon, Pennsylvania
  - GSK Investigational Site, Blue Bell, Pennsylvania
  - GSK Investigational Site, Johnstown, Pennsylvania
  - GSK Investigational Site, Latrobe, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Shippensburg, Pennsylvania
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Shelbyville, Tennessee
  - GSK Investigational Site, Allen, Texas
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Dickinson, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Gun Barrel City, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Live Oak, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sealy, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Waxahachie, Texas
  - GSK Investigational Site, Clinton, Utah
  - GSK Investigational Site, Draper, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Woods Cross, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Puyallup, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (9):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, Paraná, Entre Ríos Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Lanús
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Subiaco, Western Australia
  - GSK Investigational Site, Parkville
  - GSK Investigational Site, Randwick
- Austria (3):
  - GSK Investigational Site, Bregenz
  - GSK Investigational Site, Feldkirch
  - GSK Investigational Site, Vienna
- Belgium (5):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Gembloux
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Natoye
- Bulgaria (10):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sevlievo
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
  - GSK Investigational Site, Vidin
- Canada (5):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
- Chile (3):
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Valdivia
  - GSK Investigational Site, Viña del Mar
- GSK Investigational Site, Medellín, Colombia
- Croatia (6):
  - GSK Investigational Site, Čakovec
  - GSK Investigational Site, Dubrovnik
  - GSK Investigational Site, Jastrebarsko
  - GSK Investigational Site, Rijeka
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Česká Lípa
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- Germany (19):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Höchstadt an der Aisch, Bavaria
  - GSK Investigational Site, Weißenhorn, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Bad Pyrmont, Lower Saxony
  - GSK Investigational Site, Bad Lippspringe, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Hagen, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Telgte, North Rhine-Westphalia
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Hungary (7):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Nagykanizsa
  - GSK Investigational Site, Ráckeve
  - GSK Investigational Site, Szekszárd
  - GSK Investigational Site, Törökbálint
- Italy (8):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Sesto San Giovanni
- Latvia (2):
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Tukums
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Utena
  - GSK Investigational Site, Vilnius
- Malaysia (6):
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuching
  - GSK Investigational Site, Seremban, Negeri Sembilan
  - GSK Investigational Site, Sibu
  - GSK Investigational Site, Sungai Buloh
- Mexico (5):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Huixquilucan
  - GSK Investigational Site, Monterrey
- Peru (5):
  - GSK Investigational Site, Miraflores, Lima region
  - GSK Investigational Site, San Martín de Porres, Lima region
  - GSK Investigational Site, Santiago de Surco, Lima region
  - GSK Investigational Site, Lima
  - GSK Investigational Site, San Borja
- Philippines (4):
  - GSK Investigational Site, Dasmariñas, Cavite
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Pulilan
  - GSK Investigational Site, Quezon City
- Poland (21):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Cieszyn
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Jelenia Góra
  - GSK Investigational Site, Karpacz
  - GSK Investigational Site, Koszalin
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Sandomierz
  - GSK Investigational Site, Skarżysko-Kamienna
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zabrze
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Sibiu
- Russia (9):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- Serbia (5):
  - GSK Investigational Site, Belgrade
  - GSK Investigational Site, Čačak
  - GSK Investigational Site, Niš
  - GSK Investigational Site, Novi Sad
  - GSK Investigational Site, Užice
- Slovakia (3):
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Trnava
- South Africa (12):
  - GSK Investigational Site, Welkom, Free State
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Krugersdorp, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Thabazimbi
- South Korea (5):
  - GSK Investigational Site, Cheongju-si
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Valencia
- Taiwan (5):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (6):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Bangkoknoi
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Pathum Thani
  - GSK Investigational Site, Phitsanulok
  - GSK Investigational Site, Ratchatewi
- Ukraine (11):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kryvyi Rih
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Sumy
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Zaporizhia
- United Kingdom (19):
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Barry
  - GSK Investigational Site, Bexhill-on-Sea
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Kent
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Macclesfield
  - GSK Investigational Site, Merseyside
  - GSK Investigational Site, Penzance
  - GSK Investigational Site, Peterborough
  - GSK Investigational Site, Stockton-on-Tees
  - GSK Investigational Site, Stoke-on-Trent
  - GSK Investigational Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lee LA, Pedersen S, Pascoe SJ, Szefler SJ, Lenney W. No dose effect observed with chronic fluticasone propionate on growth velocity in children. Pediatr Allergy Immunol. 2021 Feb;32(2):377-381. doi: 10.1111/pai.13378. Epub 2020 Oct 26. No abstract available. PMID 32966707
- [Derived] Stempel DA, Szefler SJ, Pedersen S, Zeiger RS, Yeakey AM, Lee LA, Liu AH, Mitchell H, Kral KM, Raphiou IH, Prillaman BA, Buaron KS, Yun Kirby S, Pascoe SJ; VESTRI Investigators. Safety of Adding Salmeterol to Fluticasone Propionate in Children with Asthma. N Engl J Med. 2016 Sep 1;375(9):840-9. doi: 10.1056/NEJMoa1606356. PMID 27579634
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115358 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6250 participants were enrolled and randomized to study treatments; total 6208 participants took at least one dose of study drug.
Pre-assignment Details: Participants aged between 4 to 11 years having asthma, defined by the regional asthma guidelines for at least 6 months, having history of at least one occurrence of treatment with systemic corticosteroid and with no change in asthma therapy for the last 4 weeks from first visit were enrolled for the study.
Groups:
- Fluticasone Propionate/Salmeterol Combination (FSC): Participants were randomized to either FSC or FP, and the treatment dose was based on participants' asthma control status. There was no intent to compare the dosage levels received, therefore participants were combined for comparison regardless of dosage. In this treatment arm, participants received one of following treatments: FSC 100/50 microgram (µg) or FSC 250/50 µg as one inhalation twice daily (BID) (approximately 12 hours apart) via Dry powder inhaler (DPI) during the 6 month treatment period. Rescue medication (albuterol/salbutamol) via metered dose inhaler (MDI) was permitted during study treatment.
- Fluticasone Propionate (FP): Participants were randomized to either FSC or FP, and the treatment dose was based on participants' asthma control status. There was no intent to compare the dosage levels received, therefore participants were combined for comparison regardless of dosage. In this treatment arm, participants received one of the following treatments: FP 100 µg or FP 250 µg as one inhalation BID (approximately 12 hours apart) via DPI during the 6 month treatment period. Rescue medication (albuterol/salbutamol) via MDI was permitted during study treatment.
Period: Overall Study
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Started | 3107 | 3101
Completed | 2724 | 2751
Not Completed | 383 | 350
Not completed — Withdrawal by Subject | 245 | 226
Not completed — Adverse Event | 24 | 23
Not completed — Asthma Exacerbation | 34 | 35
Not completed — Lack of Efficacy | 5 | 6
Not completed — Protocol Violation | 68 | 53
Not completed — Lost to Follow-up | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- FSC DPI: Participants were randomized to either FSC or FP, and the treatment dose was based on participants' asthma control status. There was no intent to compare the dosage levels received, therefore participants were combined for comparison regardless of dosage. In this treatment arm, participants received one of following treatments: FSC 100/50 microgram (µg) or FSC 250/50 µg as one inhalation twice daily (BID) (approximately 12 hours apart) via Dry powder inhaler (DPI) during the 6 month treatment period. Rescue medication (albuterol/salbutamol) via metered dose inhaler (MDI) was permitted during study treatment.
- FP DPI: Participants were randomized to either FSC or FP, and the treatment dose was based on participants' asthma control status. There was no intent to compare the dosage levels received, therefore participants were combined for comparison regardless of dosage. In this treatment arm, participants received one of the following treatments: FP 100 µg or FP 250 µg as one inhalation BID (approximately 12 hours apart) via DPI during the 6 month treatment period. Rescue medication (albuterol/salbutamol) via MDI was permitted during study treatment.
- Total: Total of all reporting groups
Arm/Group | FSC DPI | FP DPI | Total
Number analyzed (Participants) | 3107 | 3101 | 6208
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.6 (2.21) | 7.6 (2.20) | 7.6 (2.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1187 | 1227 | 2414
  Male | 1920 | 1874 | 3794
Race/Ethnicity, Customized [Number; unit: Participants]
  African American / African Heritage | 539 | 511 | 1050
  American Indian or Alaskan Native | 144 | 118 | 262
  Asian - Central / South Asian Heritage | 30 | 37 | 67
  Asian - East Asian Heritage | 96 | 112 | 208
  Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 122 | 108 | 230
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  White - Arabic / North African Heritage | 13 | 15 | 28
  White - White / Caucasian / European Heritage | 1985 | 2017 | 4002
  Mixed Race | 167 | 180 | 347
  Missing | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Event in the Composite Safety Endpoint of Serious Asthma Outcomes ( Asthma-related Hospitalization, Asthma-related Endotracheal Intubation, or Asthma-related Death)
Description: Composite endpoint was defined as clinically relevant endpoint that is constructed from combinations of other clinically relevant endpoints of serious asthma outcomes (i.e., asthma-related hospitalization, asthma-related endotracheal intubation, or asthma-related death). Hospitalization was defined as an inpatient stay or a >=24-hour stay in an observation area in an emergency department or other equivalent facility. Time to first event in the composite endpoint of serious asthma-related outcomes over the 6-month study treatment period was analyzed using a Cox proportional hazards regression model. An estimate of absolute risk difference and its corresponding 95% confidence interval (CI) were also included. The Intent-to-Treat (ITT) Population included all participants randomized to study drug and who took study treatment.
Time Frame: From Day 1 up to 6 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 3107 | 3101
Participants | 27 | 21
Statistical Analysis 1: Comparison: FSC DPI vs FP DPI; Test type: Non-Inferiority or Equivalence — The non-inferiority comparison was statistically significant if the upper bound of the two-sided 95% CI falls below 2.675, the non-inferiority margin, and the non-inferiority test one-sided p-value <0.025; p = 0.006, Regression, Cox; Hazard Ratio (HR) = 1.285, 95% CI 2-sided [0.726 to 2.272] — Estimated for Hazard ratio
Statistical Analysis 2: Comparison: FSC DPI vs FP DPI; Test type: Superiority or Other; Risk Difference (RD) = 0.0019, 95% CI 2-sided [-0.0024 to 0.0063] — Estimated for Absolute risk difference

2. Primary Outcome: Number of Participants With at Least One Asthma Exacerbation Over the 6-month Study Treatment Period
Description: Number of participants with asthma exacerbation over the 6-month study treatment period are presented. Participants from mITT population with screening childhood asthma control test (C-ACT) scores of 20 or higher, one exacerbation in the previous year, and either low-dose inhaled corticosteroid (ICS) + one or more adjunctive therapy or medium-dose ICS monotherapy or medium-dose ICS and one or more adjunctive therapy as prior asthma therapy were included for this endpoint. Time to first exacerbation analyzed using a cox proportional hazards regression model. The number of asthma exacerbations were compared between treatments using a negative binomial regression model. The modified Intent-to-Treat (mITT) Population consisted of the ITT participants with a different data cut-off for supportive analyses of the primary composite safety endpoint.
Time Frame: From Day 1 up to 6 months
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 3107 | 3101
Participants | 265 | 309
Statistical Analysis 1: Comparison: FSC DPI vs FP DPI; Test type: Superiority or Other; Hazard Ratio (HR) = 0.859, 95% CI 2-sided [0.729 to 1.012] — Estimated for Hazard ratio

3. Secondary Outcome: Number of Participants Experiencing Asthma-related Deaths Over the 6-month Study Treatment Period.
Description: Number of participants experiencing asthma-related death over the 6-month study treatment period are presented.
Time Frame: From Day 1 up to 6 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 3107 | 3101
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing Asthma-related Endotracheal Intubations Over the 6-month Study Treatment Period
Description: Intubation is defined as endotracheal intubation with ventilation (mechanical or by hand). The number of participants experiencing asthma-related endotracheal intubations over the 6-month study treatment period are presented.
Time Frame: From Day 1 up to 6 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 3107 | 3101
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Asthma-related Hospitalizations Over the 6-month Study Treatment Period
Description: Hospitalization is defined as a >=24-hour stay as an inpatient or in an observation ward. The number of participants experiencing asthma-related hospitalizations over the 6-month study treatment period are presented.
Time Frame: From Day 1 up to 6 months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 3107 | 3101
Participants | 27 | 21

6. Secondary Outcome: Number of Participants Withdrawn From Study Treatment Due to Asthma Exacerbation Over the 6-month Study Treatment Period
Description: An exacerbation is defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days (up to 10 days) or a single depot corticosteroid injection. Number of participants experiencing at least one exacerbation from mITT population were included for this endpoint. The number of participants withdrawn from study treatment due to asthma exacerbation over the 6-month study treatment period are presented.
Time Frame: From Day 1 up to 6 months
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 265 | 309
Participants | 33 | 35

7. Secondary Outcome: Percentage of Rescue-free Days Over the 6-month Study Treatment Period
Description: Rescue-free days were days without use of rescue albuterol/salbutamol (other than pre-exercise treatment) over the 6-month study treatment period. The mean percentages of rescue-free days over the months 1-6 (defined as treatment days 2-182) are summarized. Number of participants over treatment days 2-182 from mITT Population were included for this endpoint.
Time Frame: From Day 1 up to 6 months
Population: mITT Population
Measure: Mean (Standard Error); unit: Percentage of rescue-free days
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 3049 | 3036
Percentage of rescue-free days | 83.0 (0.50) | 81.9 (0.52)

8. Secondary Outcome: Percentage of Asthma Control Days Over the 6-month Study Treatment Period
Description: An asthma control day is one on which rescue albuterol/salbutamol use was recorded as 0, no night time awakenings were recorded, no asthma exacerbations were recorded, no work, school, or daycare days were missed by caregiver or participant due to asthma, coughing symptom score was <=1 and wheezing symptom score was 0. The mean percentages of asthma control days over the months 1-6 (defined as treatment days 2-182) are summarized. Number of participants over treatment days 2-182 from mITT Population were included for this endpoint.
Time Frame: From Day 1 up to 6 months
Population: mITT Population
Measure: Mean (Standard Error); unit: Percentage of asthma control days
Arm/Group | FSC DPI | FP DPI
Number analyzed (Participants) | 2936 | 2935
Percentage of asthma control days | 74.8 (0.57) | 73.4 (0.58)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to 6 months).
Description: Due to the extensive safety database of FSC, FP, and albuterol/salbutamol, and the outcomes of interest in this study, the only non-serious AEs that were collected in this study are those that lead to study drug discontinuation.
Arm/Group | FSC DPI | FP DPI
Serious Adverse Events (participants affected / at risk) | 56/3107 | 54/3101
Other Adverse Events (participants affected / at risk) | 31/3107 | 39/3101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DPI (N=3107) | FP DPI (N=3101)
Pneumonia (Infections and infestations) | 11 | 8
Bronchitis (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bullous impetigo (Infections and infestations) | 0 | 1
Eczema infected (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pseudocroup (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral myositis (Infections and infestations) | 0 | 1
Viral tonsillitis (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 23 | 13
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 2
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Effusion (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DPI (N=3107) | FP DPI (N=3101)
Asthma (Respiratory, thoracic and mediastinal disorders) | 15 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Tremor (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Irritability (Psychiatric disorders) | 1 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Eye swelling (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.